CLINICAL TRIAL: NCT05662774
Title: The Clinical Application of Ultrasound for Acute Kidney Injury During Sepsis - From Macroscopic to Microscopic Renal Perfusion Perspectives
Brief Title: Clinical Application of Quantitative Ultrasonographic Analysis in Early Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: JD-HG-2021-40
Record Dates: First submitted 2022-11-28; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Patient Admitted to Hospital With Acute Kidney Injury Due to Sepsis
Keywords: Acute kidney injury; contrast-enhanced ultrasound; renal perfusion; microcirculation
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound contrast agent (Sonovue) — Patients are diagnosed by intravenous injection of ultrasound contrast on the first day of admission and information is collected by diagnostic ultrasound instruments

SUMMARY:
The purpose of this study was to quantify overall blood flow and renal cortical perfusion in patients with septic acute kidney injury (AKI) using ultrasound (US) Doppler and contrast-enhanced ultrasound (CEUS).

DETAILED DESCRIPTION:
Kidney ultrasound is the most widely used imaging modality in initial AKI workup as it is widely available and free of complications. It is clinically feasible to use US Doppler and contrast-enhanced US (CEUS) to detect macroscopic and microscopic changes in renal blood flow, and also cardiac output alterations.The aim was to analyze changes in US Doppler and CEUS quantitative parameters in patients with septic AKI to explore perfusion within the renal parenchyma, and also measure global renal blood flow and cardiac output.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the AKI diagnostic criteria of the Kidney Disease: Improving Global Outcomes (KDIGO)
2. Meets Sepsis 3.0 diagnostic criteria for sepsis: infection + SOFA ≥ 2

Exclusion Criteria:

1. Urinary tract obstruction, hydronephrosis, etc.
2. Left ventricular ejection fraction <30% (measured by transthoracic echocardiography), systolic pulmonary artery pressure >90 mmHg (measured by transthoracic echocardiography)
3. Allergy or adverse reaction to contrast media

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Intensive Care Unit who meet the above inclusion criteria
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Doppler parameters | First 24 hours after admission
  Time-averaged velocity (TAV)in cm/s
Ultrasound Doppler parameters | First 24 hours after admission
  Relative blood flow（RBF）in L/min
Ultrasonography parameters | First 24 hours after admission
  Time to peak (TTP)in senconds
Ultrasonography parameters | First 24 hours after admission
  Maximum intensity (Imax)in a.u（Acoustic intensity units）
Ultrasonography parameters | First 24 hours after admission
  area under curve is the multiplication of acoustic intensity and time（a.u*s）

CONTACTS AND LOCATIONS:
Overall Officials: The Second Hospital of Soochow University The Second Hospital of Soochow University, Study Chair — The Second Hospital of Soochow University
Locations (1):
- The Second Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Plan to share data publicly after patent application or academic paper publication